CLINICAL TRIAL: NCT07330570
Title: The Evaluation of Current Caries Risk in Children Treated Under General Anesthesia Due to Early Childhood Caries Between 2015-2020
Brief Title: Caries Risk in Children Treated Under General Anesthesia for Early Childhood Caries
Status: Recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Melis AKYILDIZ, Assistant Prof., Aydin Adnan Menderes University
Other Study IDs: EErsan
Record Dates: First submitted 2025-12-12; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Early Childhood Caries (ECC)
Keywords: General Anesthesia; Pediatric Dentistry; Cariogram; Caries Risk Factors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group- Children with Early Childhood Caries Treated under GA: This study includes a single group of systemically healthy children aged 6-16 years who underwent dental treatment under general anesthesia for early childhood caries (ECC) between 2015 and 2020 at Aydın Adnan Menderes University Faculty of Dentistry.
  Interventions: Diagnostic Test: Caries Risk Assesment

INTERVENTIONS:
Diagnostic Test: Caries Risk Assesment — Participants will undergo a single-visit evaluation in which caries risk will be comprehensively assessed using the Cariogram model. The assessment will integrate findings from clinical examination (including DMFT/dmft scores, Plaque Index, Gingival Index, and probing depth), salivary analysis (stimulated flow rate and buffer capacity), and standardized questionnaires evaluating diet, fluoride exposure, socioeconomic status, and dental visit history. No treatment or experimental intervention will be performed; all data will be collected exclusively for observational analysis.

SUMMARY:
This observational, cross-sectional study aims to evaluate the current caries risk profiles of children who underwent dental treatment under general anesthesia (GA) for early childhood caries (ECC) between 2015 and 2020 at Aydın Adnan Menderes University, Faculty of Dentistry. A minimum of 44 systemically healthy children will be included.

Caries risk will be assessed using the Cariogram model, incorporating clinical parameters (DMFT/dmft, Plaque Index, Gingival Index, probing depth), salivary factors (stimulated flow rate, buffer capacity), and standardized questionnaires covering diet, fluoride exposure, socioeconomic status, and dental visit history. Data will be collected in a single visit, analyzed using SPSS.

The study aims to provide scientific evidence for long-term preventive strategies and oral health policies targeting high-risk pediatric populations treated under GA for ECC.

DETAILED DESCRIPTION:
Early childhood caries (ECC) is defined as the presence of one or more decayed, missing, or filled primary teeth in children, particularly those aged 71 months or younger. ECC is one of the most common chronic diseases of childhood, with a prevalence reaching up to 70% in communities with low socioeconomic status. According to the data from the Turkish Oral and Dental Health Profile studies, while a decrease in the average number of decayed teeth and dmft index was observed in 2018 compared to 2004, an increase in the average number of filled and missing teeth was detected. Although this demonstrates improved access to caries treatment services, the persistently high prevalence of ECC indicates a continuing need for effective preventive strategies.

In the treatment of ECC, particularly in younger children with extensive caries and challenging behavior management, dental interventions are frequently performed under general anesthesia (GA). However, long-term follow-up studies have shown insufficient attention to oral hygiene and limited access to preventive applications among children treated under GA. Research on this patient group reveals a high incidence of recurrent caries after treatment. These findings indicate that approaches focusing solely on treatment are insufficient, as the risk of caries persists, and these individuals require long-term, structured follow-up.

The aim of this thesis study is to objectively evaluate the current caries risk levels of individuals who underwent dental treatment under GA for ECC. For this purpose, children treated for ECC under GA at Aydın Adnan Menderes University Faculty of Dentistry between 2015 and 2020 will be recalled, and their current caries risk profiles will be analyzed using the Cariogram model, the most up-to-date official web-based version available at "cariogram.uni.mau.se".

Caries risk assessment will be performed using a comprehensive set of parameters integrated into the Cariogram model, including:

* Clinical caries experience (DMFT/dmft indices),
* Oral hygiene status (Plaque Index, Gingival Index, probing depth),
* Salivary factors (stimulated flow rate, buffer capacity,)
* Diet content and frequency,
* Fluoride exposure,
* Socioeconomic status,
* Past dental history and frequency of dental visits,
* General health and medication use.

Each parameter will be scored according to standardized criteria. Participants will be invited only once, and the study will have a cross-sectional design, with data collection completed in a single visit.

This research will provide scientific data for monitoring and protecting high-risk pediatric populations at both individual and community levels in the fight against caries. Furthermore, the findings are expected to contribute to the planning of preventive oral health services and the development of oral health policies. By examining the course of caries risk in individuals treated under GA for ECC in later years, this study will help better understand the need for preventive care in this population. These evaluations will not only reveal the current situation but also contribute to the development of effective and sustainable preventive service models for these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who underwent dental treatment under general anesthesia for early childhood caries (ECC) at the Department of Pediatric Dentistry, Faculty of Dentistry, Aydın Adnan Menderes University between 2015-2020
* Patients whose follow-up information (e.g., discharge summary, treatment plan) is accessible through clinical records
* Individuals who provide written informed consent signed by their parents/legal guardians and assent from the child to participate in the study

Exclusion Criteria:

* Individuals with medical conditions that may affect oral health, such as systemic diseases, immunodeficiencies, or chronic illnesses
* Children with special healthcare needs or mental/physical disabilities
* Patients who do not cooperate during the examination or do not allow the completion of the oral examination

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 6-16 years who underwent dental treatment under general anesthesia for early childhood caries (ECC) at Aydın Adnan Menderes University, Faculty of Dentistry between 2015-2020
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Caries Risk Assessment | Baseline
  Caries risk will be evaluated using the Cariogram model, which combines clinical, salivary, behavioral, and socioeconomic factors to estimate each participant's "chance to avoid caries." Key inputs include caries experience (DMFT/dmft), plaque and gingival status, salivary flow and buffering, diet and oral hygiene habits, fluoride exposure, dental attendance, and socioeconomic or health-related influences. The Cariogram software will integrate these variables to generate a visual risk profile and a final percentage score for objective comparison between participants. The following parameters are evaluated in the Cariogram:
  Caries History Systemic disease: 0: No disease, 1: a mild systemic disease, 2: Severely affecting systemic diseaseDietary content: the cariogenic potential of foods 0: ≤ 10³ CFU/ml, 1: 10⁴ CFU/ ml, 2: 10⁵ CFU/ml, 3: ≥10⁶ CFU/ml Diet frequency: Average daily number of meals and snacks 0≤ 3 meals/day, 1: 4-5 meals/day, 2: 6-7 meals/day, 3: >7 meals/day

SECONDARY OUTCOMES:
DMFT/dmft Scores | Baseline
  DMFT/dfs index in individuals consists of the following components:
  D (Decayed): Number of decayed and untreated permanent teeth M (Missing): Number of permanent teeth extracted due to caries F (Filled): Number of permanent teeth restored with fillings T(Teeth) For each participant, these three components will be recorded separately, and the total DMFT score will be calculated.
  0: DMFT=0, 1: DMFT=1, 2: DMFT=2, 3: DMFT ≥ 3
Plaque Index (Silness-Löe) | Baseline
  Oral hygiene status will be assessed using the standardized Plaque Index criteria on specified tooth surfaces. Plaque Index (PI) - Silness and Löe 0: No plaque
  1. Thin visible plaque, difficult to detect
  2. Thick visible plaque, easily detectable
  3. Presence of plaque filling the interproximal area
  0: 0 (Excellent), 1: 0.1-0.9 (Good), 2: 1.0-1.9 (Moderate), 3: 2.0-3.0 (Poor)
Gingival Index (Löe-Silness) | Baseline
  Gingival health will be measured using the Gingival Index to evaluate the degree of gingival inflammation.
  0: Normal gingiva - no edema, 1: Mild edema, no bleeding after gentle probing, 2: Moderate to severe gingival edema, bleeding after air drying, 3: Severe inflammation; redness and edema. Ulceration. Tendency for spontaneous bleeding
Stimulated Salivary Flow Rate (mL/min) | Baseline
  Stimulated salivary flow rate will be measured using wax-stimulated saliva collection and expressed in mL/min.
  0: ≥0.7 mL/min
  1. 0.3-0.7 mL/min
  2. <0.3 mL/min
Salivary Buffering Capacity (pH) | Baseline
  Salivary buffering capacity will be assessed using Dentobuff test strips to measure salivary pH.
  0: pH ≥6.0
  1. pH 4.5-5.5
  2. pH ≤4.0
Probing Depth (mm) | Baseline
  Probing depth refers to the distance (in millimeters) between the gingival margin and the deepest point of the periodontal tissues surrounding the tooth that can be probed. This measurement is performed using a special instrument called a periodontal probe, which has a rounded tip and is calibrated in millimeters.
  1-3 mm: Healthy gingiva/sulcus, 4 mm: Initial periodontal disease, 5-6 mm: Moderate periodontitis, ≥7 mm: Advanced periodontitis
Fluoride Program | Baseline
  The amount of fluoride present in the mouth. Obtained through interview. 0: Maximum Program, 1: Supplement, 2: Toothpaste Only, 3: No Fluoride

CONTACTS AND LOCATIONS:
Overall Officials: Melis Akyıldız, Principal Investigator — Aydın Adnan Menderes University, Faculty of Dentistry
Locations (1):
- Aydın Adnan Menderes University, Faculty of Dentistry, Aydin, Aydın, Turkey (Türkiye)

REFERENCES:
- [Background] American Academy of Pediatric Dentistry. (2023). Definition of Early Childhood Caries (ECC). AAPD Reference Manual.
- [Background] Kirthiga M, Murugan M, Saikia A, Kirubakaran R. Risk Factors for Early Childhood Caries: A Systematic Review and Meta-Analysis of Case Control and Cohort Studies. Pediatr Dent. 2019 Mar 15;41(2):95-112. PMID 30992106
- [Background] T.C. Sağlık Bakanlığı. (2004). Türkiye Ağız ve Diş Sağlığı Profili (TADSAP-2004). Refik Saydam Hıfzıssıhha Merkezi Başkanlığı Yayınları.
- [Background] T.C. Sağlık Bakanlığı. (2018). Türkiye Ağız ve Diş Sağlığı Profili (TADSAP-2018). Türkiye Halk Sağlığı Kurumu Yayınları.
- [Background] Casamassimo PS, Thikkurissy S, Edelstein BL, Maiorini E. Beyond the dmft: the human and economic cost of early childhood caries. J Am Dent Assoc. 2009 Jun;140(6):650-7. doi: 10.14219/jada.archive.2009.0250. PMID 19491160
- [Background] Kim Seow W. Environmental, maternal, and child factors which contribute to early childhood caries: a unifying conceptual model. Int J Paediatr Dent. 2012 May;22(3):157-68. doi: 10.1111/j.1365-263X.2011.01186.x. Epub 2011 Oct 4. PMID 21972925
- [Background] Oubenyahya H, Bouhabba N. General anesthesia in the management of early childhood caries: an overview. J Dent Anesth Pain Med. 2019 Dec;19(6):313-322. doi: 10.17245/jdapm.2019.19.6.313. Epub 2019 Dec 27. PMID 31942447
- [Background] Williams C, Kendall L. Tackling strokes. Nurs Times. 1998 Aug 12-18;94(32):32-3. PMID 9752176
- [Background] Li JY, He SY, Wang PX, Dai SS, Zhang SQ, Li ZY, Guo QY, Liu F. Incidence and risk factors of unplanned retreatment following dental general anesthesia in children with severe early childhood caries. Front Pediatr. 2023 Jul 27;11:1163368. doi: 10.3389/fped.2023.1163368. eCollection 2023. PMID 37576136
- [Background] Featherstone JD. The continuum of dental caries--evidence for a dynamic disease process. J Dent Res. 2004;83 Spec No C:C39-42. doi: 10.1177/154405910408301s08. PMID 15286120
- [Background] Bratthall D, Hansel Petersson G. Cariogram--a multifactorial risk assessment model for a multifactorial disease. Community Dent Oral Epidemiol. 2005 Aug;33(4):256-64. doi: 10.1111/j.1600-0528.2005.00233.x. PMID 16008632
- [Background] Twetman S, Fontana M, Featherstone JD. Risk assessment - can we achieve consensus? Community Dent Oral Epidemiol. 2013 Feb;41(1):e64-70. doi: 10.1111/cdoe.12026. PMID 24916679
- [Background] Taqi M, Zaidi SJA. Predictive validity of the reduced Cariogram model for caries increment in non-cavitated and cavitated lesions: cohort study. BMC Oral Health. 2023 Oct 24;23(1):790. doi: 10.1186/s12903-023-03479-w. PMID 37875839
- [Background] Gao XL, Hsu CY, Xu Y, Hwarng HB, Loh T, Koh D. Building caries risk assessment models for children. J Dent Res. 2010 Jun;89(6):637-43. doi: 10.1177/0022034510364489. Epub 2010 Apr 16. PMID 20400721
- [Background] Campus G, Cagetti MG, Sale S, Carta G, Lingstrom P. Cariogram validity in schoolchildren: a two-year follow-up study. Caries Res. 2012;46(1):16-22. doi: 10.1159/000334932. Epub 2012 Jan 4. PMID 22222621
- [Background] Utreja, D., Singh, A., Purohit, B. M., & Purohit, R. N. (2019). Application of Cariogram in Caries Risk Assessment Among Schoolchildren in India. Oral Health & Preventive Dentistry, 17(2), 133-138
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Al Shayeb KN, Turner W, Gillam DG. Periodontal probing: a review. Prim Dent J. 2014 Aug;3(3):25-9. doi: 10.1308/205016814812736619. PMID 25198634
- [Background] Gugnani N, Pandit IK, Srivastava N, Gupta M, Sharma M. International Caries Detection and Assessment System (ICDAS): A New Concept. Int J Clin Pediatr Dent. 2011 May-Aug;4(2):93-100. doi: 10.5005/jp-journals-10005-1089. Epub 2010 Apr 15. PMID 27672245
- [Background] Cavalcante, G. M. S., Teles, R. P., Scarparo, R. K., Silva, M. E. R., & Mialhe, F. L. (2014). Dental caries experience among children with cerebral palsy in Brazil: A case-control study. Journal of Applied Oral Science, 22(3), 215-220. https://doi.org/10.1590/1678-775720130689